CLINICAL TRIAL: NCT03942029
Title: Safety and Tolerability of LY3154207 in Combination With a CYP3A4 Inhibitor and Assessment of Pharmacokinetics of LY3154207 After Administration of Capsule and Tablet Formulations in Healthy Subjects
Brief Title: A Drug Interaction Study of LY3154207 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 16304; I7S-MC-HBEF (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01-15

CONDITIONS: Healthy
MeSH Terms: interventions — LY3154207; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The capsule versus tablet formulation comparison will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 Part A - LY3154207 Capsule (Experimental): LY3154207 capsule (reference) administered orally, once.
  Interventions: Drug: LY3154207 Capsule
- Cohort 1 Part A - LY3154207 Tablet (Experimental): LY3154207 tablet (test) administered orally, once.
  Interventions: Drug: LY3154207 Tablet
- Cohort 1 Part B LY3154207 (Dose 1) + Fluconazole (Experimental): LY3154207 (dose 1) administered alone, orally once. Fluconazole administered alone, orally, on consecutive days. LY3154207 co-administered with fluconazole on consecutive days.
  Interventions: Drug: LY3154207 Tablet; Drug: Fluconazole Tablet
- Cohort 1 Part B - Placebo + Fluconazole (Experimental): Placebo administered alone, orally, once. Fluconazole administered alone, orally, on consecutive days. Placebo co-administered with fluconazole on consecutive days.
  Interventions: Drug: Placebo; Drug: Fluconazole Tablet
- Cohort 2 - LY3154207 (Dose 2) + Fluconazole (Experimental): LY3154207 (dose 2) administered alone, orally once. Fluconazole administered alone, orally, on consecutive days. LY3154207 co-administered with fluconazole on consecutive days.
  Interventions: Drug: LY3154207 Tablet; Drug: Fluconazole Tablet
- Cohort 2 - Placebo + Fluconazole (Experimental): Placebo administered alone, orally once. Fluconazole administered alone, orally, on consecutive days. Placebo co-administered with fluconazole on consecutive days.
  Interventions: Drug: Placebo; Drug: Fluconazole Tablet
- Cohort 3 - LY3154207 + Fluconazole (Experimental): LY3154207 (dose 2) administered alone, orally, on consecutive days. LY3154207 co-administered with fluconazole on consecutive days.
  Interventions: Drug: LY3154207 Tablet; Drug: Fluconazole Tablet
- Cohort 3 - Placebo + Fluconazole (Experimental): Placebo administered alone, orally, on consecutive days. Placebo co-administered with fluconazole on consecutive days.
  Interventions: Drug: Placebo; Drug: Fluconazole Tablet

INTERVENTIONS:
Drug: LY3154207 Capsule — Administered orally as capsule
  Arms: Cohort 1 Part A - LY3154207 Capsule
Drug: LY3154207 Tablet — Administered orally as tablet
  Arms: Cohort 1 Part A - LY3154207 Tablet; Cohort 1 Part B LY3154207 (Dose 1) + Fluconazole; Cohort 2 - LY3154207 (Dose 2) + Fluconazole; Cohort 3 - LY3154207 + Fluconazole
Drug: Placebo — Administered orally as tablet
  Other Names: Placebo Tablet
  Arms: Cohort 1 Part B - Placebo + Fluconazole; Cohort 2 - Placebo + Fluconazole; Cohort 3 - Placebo + Fluconazole
Drug: Fluconazole Tablet — Administered orally as tablet
  Arms: Cohort 1 Part B - Placebo + Fluconazole; Cohort 1 Part B LY3154207 (Dose 1) + Fluconazole; Cohort 2 - LY3154207 (Dose 2) + Fluconazole; Cohort 2 - Placebo + Fluconazole; Cohort 3 - LY3154207 + Fluconazole; Cohort 3 - Placebo + Fluconazole

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of LY3154207 and fluconazole (anti-fungal medication), when taken together by healthy participants. The study will last from nine to 11 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 18 to 35 kilogram per meter square (kg/m²)
* Have clinical laboratory test results within acceptable range for the population

Exclusion Criteria:

* Have consumed grapefruits or grapefruit-containing products, Seville oranges or Seville orange-containing products, star fruits or star fruit-containing products within 7 days prior to dosing or intend to consume during the study
* Intend to use over-the-counter or prescription medication (with exception of hormonal contraceptives and acetaminophen), including herbal preparations containing St. John's wort, kava, garlic, ginger, ginkgo biloba, or guarana, within 14 days prior to Check-in and during the study
* Use of any drugs or substances that are known inducers and/or inhibitors of cytochrome P450 (CYP) 3A within 14 days prior to the administration of study drug and during the study
* Have evidence of active renal disease (eg, diabetic renal disease, polycystic kidney disease) or an estimated creatinine clearance of < 80 milliliters per minute (mL/minute), calculated using the Chronic Kidney Disease Epidemiology Collaboration equation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline up to 11 weeks
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Change from Baseline in Blood Pressure (BP) | Baseline, up to 48 hours post dose when LY3154207 is co-administered with fluconazole
  BP measured by ambulatory blood pressure monitoring (ABPM)
Change from Baseline in Pulse Rate (PR) | Baseline, up to 48 hours post dose when LY3154207 is co-administered with fluconazole
  PR measured by ABPM
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3154207 | Baseline up to 48 hours postdose
  PK: Cmax of LY3154207
PK: Area Under the Concentration Versus Time Curve from Time Zero to Time T, where T is the Last Sample with a Measurable Concentration (AUC[0-tlast]) of LY3154207 | Baseline up to 48 hours postdose
  PK: AUC(0-tlast) of LY3154207
PK: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf]) of LY3154207 | Baseline up to 48 hours postdose
  PK: AUC(0-inf) of LY3154207

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No